CLINICAL TRIAL: NCT02487485
Title: Examining the Impact of Sirolimus on Ketamine's Antidepressant Effects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 1504015604
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Ketamine; Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketamine + sirolimus (placebo at time 2) (Experimental): Participants will be treated twice with ketamine 0.5 mg/kg infused over 40 minutes, combined with a single dose of sirolimus 6 mg orally. After two weeks, they will recieve another infusion of ketamine, and a single dose of placebo.
  Interventions: Drug: Ketamine; Drug: sirolimus; Drug: Placebo
- ketamine + placebo (sirolimus at time 2) (Placebo Comparator): Participants will be treated twice with ketamine 0.5 mg/kg infused over 40 minutes, combined with a single dose of sirolimus 6 mg placebo. After two weeks, they will recieve another infusion of ketamine, and a single dose of sirolimus 6 mg.
  Interventions: Drug: Ketamine; Drug: sirolimus; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — . Subjects will receive an infusion of ketamine (0.5 mg/kg infusion over approximately 40 minutes). All subjects will receive two ketamine infusions-once with a placebo and once with a single dose of sirolimus (6 mg, oral administration).
Drug: sirolimus — Subjects will receive a single 6 mg oral dose via oral solution of sirolimus or a dose of placebo approximately two hours prior to the infusions. As above, the order of placebo and sirolimus is randomized. The sirolimus dose as well as the placebo solution will be given in 6 ounces of orange juice.
  Other Names: Rapamune
Drug: Placebo — Placebo oral dose

SUMMARY:
The aim of the study is to provide insight into the impact of the immunosuppressant drug sirolimus, on the antidepressant effects of the prototypal rapid-acting antidepressant medication, ketamine.

DETAILED DESCRIPTION:
This is a double blind, placebo-controlled, crossover, randomized controlled trial investigating the impact of sirolimus on ketamine's antidepressant effects in participants with antidepressant-resistant depressive symptoms.

Prior to this, there was a phase 1 which included monitoring 3 subjects over the course of 7 days after a single dose of sirolimus and ketamine in order to inquire about side effects or interaction effects.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans and non-Veterans between the ages of 21-65.
2. Diagnosis of Major Depressive Episode (unipolar or bipolar) as determined by the Mini International Neuropsychiatric Interview (MINI).
3. Antidepressant-resistant depressive symptoms, defined by a history of failure of one or more adequate antidepressant trials.
4. Stable doses of antidepressants (if prescribed) for a period of four weeks or longer at the time of randomization, except for MAOIs which are prohibited.
5. Stable course of psychotherapy (if engaged in) for a period of four weeks or longer at the time of randomization.
6. Females will be included if they are not pregnant or breastfeeding and agree to utilize a medically accepted birth control method (to include oral, injectable, or implant birth control, condom, diaphragm with spermicide, intrauterine device, tubal ligation, abstinence, or partner with vasectomy) or if post-menopausal for at least 1 year, or surgically sterile. For those women who are taking an oral contraceptive, we will also ask that they use (or ask their partners to use) a barrier method contraceptive.
7. Able to provide written informed consent according to VA HSS guidelines.
8. Ability to read and write in English.
9. A score greater than or equal to 18 on the Montgomery Åsberg Depression Rating Scale (MADRS).

Exclusion Criteria:

1. Subjects with a diagnostic history of schizophrenia or schizoaffective disorder, or currently exhibiting manic or mixed episodes or psychotic features as confirmed by the Mini International Neuropsychiatric Inventory.
2. Current, ongoing serious suicidal risk as assessed by evaluating investigator or by scoring 5 or more on the item-10 of the MADRS.
3. Patients with unstable or inadequately controlled medical conditions.
4. Patient requiring prohibited medication.
5. Patient with history of organ transplant.
6. Meet criteria for a diagnosis of substance dependence (amphetamines, cocaine, hallucinogens, inhalants, opioids, sedatives/hypnotics/anxiolytics) within the three months prior to screening date.
7. Positive urine drug screen for cannabis, cocaine, PCP, or barbiturates.
8. Positive pregnancy test at screening at any screen given during the study.
9. Known sensitivity to sirolimus or ketamine.
10. History of sensitivity to heparin or heparin-induced thrombocytopenia.
11. Resting blood pressure lower than 85/55 or higher than 150/95, or resting heart rate lower than 45/min or higher than 100/min.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Abdallah, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - West Haven Veterans Affairs, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine + Sirolimus First, Then Ketamine + Placebo: Participants received ketamine 0.5 mg/kg infused over 40 minutes, combined with a single dose of sirolimus 6 mg orally. After two weeks, they received another infusion of ketamine, and a single dose of placebo.
- Ketamine + Placebo First, Then Ketamine + Sirolimus: Participants received ketamine 0.5 mg/kg infused over 40 minutes, combined with a single dose of placebo. After two weeks, they received another infusion of ketamine, and a single dose of sirolimus 6 mg.
Period: Overall Study
Arm/Group | Ketamine + Sirolimus First, Then Ketamine + Placebo | Ketamine + Placebo First, Then Ketamine + Sirolimus
Started | 12 | 11
Completed | 9 | 8
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine + Sirolimus First, Then Ketamine + Placebo | Ketamine + Placebo First, Then Ketamine + Sirolimus | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.09 (13.22) | 44.1 (12.6) | 42 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Montgomery-Asberg Depression Rating Scale (MADRS): The MADRS is a standardized instrument to ascertain depressed mood and neurovegetative signs and symptoms of depression. Ranges from 0-60 (higher is worse).
Time Frame: Pretreatment and 2 week
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Ketamine + Sirolimus: Participants received ketamine 0.5 mg/kg infused over 40 minutes, combined with a single dose of sirolimus 6 mg orally.
- Ketamine + Placebo: Participants received ketamine 0.5 mg/kg infused over 40 minutes, combined with a single dose of placebo.
Arm/Group | Ketamine + Sirolimus | Ketamine + Placebo
Number analyzed (Participants) | 20 | 20
score on a scale
  Pretreatment | 27.9387 (1.9) | 26.5756 (1.9)
  At 2 weeks | 16.5482 (2.3) | 20.9065 (2.3)

2. Secondary Outcome: Quick Inventory of Depressive Symptoms (QIDS)
Description: Quick Inventory of Depressive Symptoms - Self-Report (QIDS-SR): The QIDS-SR is a patient-rated depression instrument. Ranges from 0-27 (higher is worse).
Time Frame: Pretreatment and 2 week
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ketamine + Sirolimus | Ketamine + Placebo
Number analyzed (Participants) | 20 | 20
score on a scale
  Pretreatment | 12.6342 (1.4) | 11.3942 (1.4)
  At 2 weeks | 9.1193 (1.2) | 10.6699 (1.3)

3. Secondary Outcome: Hamilton Anxiety Rating Scale (HAMA)
Description: Hamilton Anxiety Rating Scale (HAM-A): The HAM-A is a standardized clinician-rated instrument to evaluate the severity of anxiety symptoms. Ranges from 0-56 (higher is worse).
Time Frame: Pretreatment and 2 week
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ketamine + Sirolimus | Ketamine + Placebo
Number analyzed (Participants) | 20 | 20
score on a scale
  Pretreatment | 12.9678 (1.4) | 13.8222 (1.4)
  At 2 weeks | 9.8755 (1.4) | 10.8669 (1.6)

4. Secondary Outcome: Clinician Administered Dissociative States Scale (CADSS)
Description: Clinician Administered Dissociative States Scale (CADSS): The CADSS has self and interviewer-administered items including 5 subscales, generated a priori, evaluating dissociation including altered environmental perception, time perception, spatial/body perception, derealization and memory impairment. Ranges from 0-108 (higher is worse).
Time Frame: During infusion, approximately 40 mins
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ketamine + Sirolimus | Ketamine + Placebo
Number analyzed (Participants) | 20 | 20
score on a scale | 12.1 (3.1) | 13.95 (3.1)

5. Secondary Outcome: Positive and Negative Symptom Scale (PANSS) - Positive
Description: Positive and Negative Symptom Scale (PANSS): The PANSS is commonly used to measure the severity of symptoms in psychotic disorders. It is a clinician- administered scale and includes three categories of symptoms: (1) positive symptoms, such as hallucination and delusion; (2) negative symptoms, such as flat affect and difficulty in abstract thinking; (3) general psychopathology, such as mannerisms and posturing. Ranges from 0-49 for positive scale (higher is worse).
Time Frame: During infusion, approximately 40 mins
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ketamine + Sirolimus | Ketamine + Placebo
Number analyzed (Participants) | 20 | 20
score on a scale | 9.1537 (0.59) | 8.9444 (0.60)

6. Secondary Outcome: Rapamycin Level
Description: Plasma level of rapamycin (a.k.a. sirolimus).
Time Frame: During infusion, approximately 0 mins
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Ketamine + Sirolimus | Ketamine + Placebo
Number analyzed (Participants) | 20 | 20
ng/mL | 26.5 (2.4) | 0 (0)

7. Secondary Outcome: Ketamine Level
Description: Plasma level of ketamine
Time Frame: During infusion, approximately 40 mins
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Ketamine + Sirolimus | Ketamine + Placebo
Number analyzed (Participants) | 20 | 20
ng/mL | 115 (16) | 125 (13)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Ketamine + Sirolimus | Ketamine + Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine + Sirolimus (N=20) | Ketamine + Placebo (N=20)
Anxiety (Psychiatric disorders) | 1 | 0 (0)
Chest Tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Dizzy (General disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dry Mouth (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 3
Fever (General disorders) | 1 | 0
GI Discomfort (Gastrointestinal disorders) | 2 | 0
Headaches (Nervous system disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 3 | 2
Pain (General disorders) | 3 | 1
Upper Respiratory Issues (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT02487485/Prot_SAP_000.pdf